CLINICAL TRIAL: NCT01621386
Title: A Study Comparing Measures of Ventilatory Heterogeneity (VH) in Asthma Patients
Brief Title: Ventilatory Heterogeneity in Participants With Asthma (MK-0476-513)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hal C Charles (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Hal C Charles, Associate Professor, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00038169; MK-0476-513 (Other: Merck Protocol Number)
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Participants (Experimental): Participants (male or female) that are between 18-65 years of age with a clinical diagnosis of asthma will take montelukast for 2 weeks (treatment period 1) and then take prednisone for 2 weeks (treatment period 2)
  Interventions: Drug: Montelukast; Drug: Prednisone

INTERVENTIONS:
Drug: Montelukast — Administered orally as a single daily 10 mg dose for 2 weeks
  Other Names: Singulair
Drug: Prednisone — Administered orally as a single daily 20 mg dose for 2 weeks

SUMMARY:
This study will explore the utility of magnetic resonance imaging (MRI) to assess ventilatory defects that occur due to asthma, determine the sensitivity and specificity of MRI in response to drug treatment, and whether MRI can serve as a biomarker of treatment effects due to asthma therapy.

ELIGIBILITY:
Inclusion Criteria (ALL Patients)

* Patient is a male or female 18 to 65 years of age with clinical diagnosis of asthma for at least 1 year at the prestudy (screening) visit.
* For female patients of reproductive potential, a blood pregnancy test will be performed, and it must be negative before the patient can continue in this study. If sexually active, the patient must agree to use appropriate contraceptive measures for the duration of the study and for 2 weeks after Visit 5. Medically acceptable contraceptives include: (1) surgical sterilization (such as a tubal ligation or hysterectomy), (2) approved hormonal contraceptives (such as birth control pills, patches, implants or injections), (3) barrier methods (such as a condom or diaphragm) used with a spermicide, or (4) an intrauterine device (IUD). Contraceptive measures such as Plan B™, sold for emergency use after unprotected sex, are not acceptable methods for routine use.
* Patient understands the study procedures and agrees to participate in the study by giving written informed consent (Consent must be given before any study procedures are performed)
* Patient is willing to comply with the study restrictions and adhere to the visit/protocol schedules.
* Patient is judged to be in good health (except for asthma) based on medical history, physical examination, vital sign measurements, and laboratory safety tests performed at the prestudy (screening) visit and/or prior to administration of the initial dose of study drug and has no evidence of cardiac, endocrine, or metabolic disease.
* Patient has a Body Mass Index (BMI) ≤ 39 kg/m2 at the prestudy screening (Visit 1). BMI is calculated by taking the patient's weight in kg and dividing by the patient's height in meters, squared. Patient's body must fit within the scanner sufficiently well to allow satisfactory imaging in the opinion of the investigator.
* Patient is a current non-smoker or if patient has a history of smoking, has not smoked for at least 6 months and has a smoking history of no more than 5 pack-years (i.e., 1 pack per day for 5 years). Patients who have discontinued smoking or the use of nicotine / nicotine containing products for at least approximately 3 months may be enrolled in the study at the discretion of the investigator.
* Patient has been defined by the study site team as having allergic asthma.
* Patient is able to perform reproducible pulmonary function testing (i.e., the 2 best acceptable spirograms have FEV1 values that do not vary by more than 5% of the largest value or more than 100 mL, whichever is greater).
* Patient has no clinically significant abnormality on electrocardiogram (ECG) performed at the prestudy (screening) visit and/or prior to administration of the initial dose of study drug.
* Patient has no contraindication to MRI exam.

Additional Inclusion Criteria- Mild Asthma

* Known diagnosis of asthma for at least one year as defined by NHLBI NAEPP guidelines. (http://www.nhlbi.nih.gov/guidelines/asthma/execsumm.pdf).
* FEV1 > 80% predicted
* Either reversibility of airflow obstruction after 4 puffs inhaled albuterol of 12% in either the FEV1 or FVC, or hyperresponsiveness by methacholine with PC20 FEV1 < 16 mg/ml.
* Asthma Control Questionnaire score < 1.25 consistent with good control

Additional Inclusion Criteria- Moderate and Severe Asthma

- Known diagnosis of asthma for at least one year as defined by NHLBI NAEPP guidelines. (http://www.nhlbi.nih.gov/guidelines/asthma/execsumm.pdf).

MODERATE:

* Symptoms consistent with moderate asthma as defined by 2007 NAEPP guidelines.
* Treatment with low to medium dose ICS +/- a second controller (long acting beta agonist but not leukotriene antagonist).
* Spirometry consistent with moderate asthma as defined by NHLBI NAEPP guidelines and evidence of either reversibility of airflow obstruction after 4 puffs inhaled albuterol of 12% in either the FEV1 or FVC, or hyperresponsiveness by methacholine with PC20 FEV1 < 16 mg/ml.

SEVERE:

* Treatment with high dose inhaled corticosteroids equivalent to fluticasone > 880 μg/day or beclomethasone > 1260 μg/day.
* Two of the Following:

  1. Requirement for daily controller therapy in addition to inhaled corticosteroids including long acting beta agonist but not leukotriene antagonist
  2. Symptoms requiring short acting beta agonist use daily
  3. Persistent airway obstruction (FEV1 < 80%, peak expiratory flow variability > 20%)
  4. One or more urgent care visits for asthma per year
  5. Three or more "bursts" of oral corticosteroids per year
  6. Prompt deterioration with greater than 25% reduction in inhaled or oral corticosteroid dose

Note: near fatal asthma event in the past is part of the definition, but subjects will not be eligible for study if they fulfill this criterion within the past 5 years.

Exclusion Criteria

* Patient is mentally or legally incapacitated, has significant emotional problems at the time of Screening (Visit 1) or expected during the conduct of the study or has a history of a clinically significant psychiatric disorder over the last 5 years. Subjects who have had situational depression may be enrolled in the study at the discretion of the investigator.
* Patient has taken an investigational product within 4 weeks prior to the prestudy (screening) visit. The 4 week window will be derived from the date of the last dose of study drug in the previous study to the prestudy/screening visit of the current study.
* Patient has a history of any illness that, in the opinion of the study investigator, might confound the results of the study or poses an additional risk to the subject by their participation in the study including, but not limited to, diabetes mellitus, hypertension, osteoporosis, as well as poorly controlled concomitant conditions that include obstructive sleep apnea (OSA), gastroesophageal reflux disease (GERD), and chronic sinusitis/rhinitis.
* Students or employees who are under direct supervision by any of the investigators in this protocol are not eligible to participate.
* Patient has significant or unexplained abnormalities on the physical examination and/or laboratory safety tests at Visit 1.
* Patient has a blood pressure of >150 mm Hg systolic or >95 mm Hg diastolic on >2 measurements done >5 minutes apart at Visit 1 or Visit 2.
* Patient has ECG abnormalities consistent with previous myocardial infarction, hypertrophic cardiomyopathy, ischemic heart disease or conduction system disease.
* Patient has evidence of illness that would require treatment with an excluded medication, could be immediately life threatening (e.g., arrhythmias, congenital heart disease), would pose a restriction on participation or successful completion of the study, or would pose an additional risk to administering montelukast to the patient.
* History of intubation due to asthma within the last five (5) years.
* FEV1 < 45% predicted
* Hospitalization within previous 6 months
* Patient has had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 8 weeks prior to the prestudy (screening) visit.

  m. Patient has a history of significant multiple and/or severe allergies to medications used (or potentially used) in this study (including albuterol, montelukast, prednisone, acetaminophen, lidocaine, fentanyl, atropine, and midazolam as well as latex), or has had an anaphylactic reaction or significant intolerability to a marketed or investigational prescription or non-prescription drug or to food.
* Patient has a history of stroke, chronic seizures, or major neurological disorder.
* Patient has a history of neoplastic disease.
* Patient is a female who is ≤8 weeks postpartum or breast feeding an infant.
* Patient is pregnant as determined by initial serum β-HCG obtained at Visit 1, becomes pregnant during the study as determined by urine pregnancy testing during subsequent Visits (#2-5), or intends to become pregnant during the time course of the study.
* Patient has an implanted mechanically, electrically or magnetically activated device or any metal in their body which cannot be removed, including but not limited to: pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bioprosthesis, artificial limb, metallic fragment or foreign body, shunt, surgical staples (including clips or metallic sutures) and/or ear implants.
* Patient is unable to perform breath holding or spirometry maneuvers or to tolerate immobilization within the MRI scanner.
* Patient consumes excessive amounts of alcohol, defined as greater than 3 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [284 mL/10 ounces], wine [125 mL/4 ounces], or distilled spirits [25 mL/1 ounce]) per day. Subjects that consume 4 glasses of alcoholic beverages per day may be enrolled at the discretion of the investigator.
* Patient consumes excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, or other caffeinated beverages per day.
* Patient is currently a regular user (including "recreational use") of any illicit drugs or has a history of drug (including alcohol) abuse within approximately 12 months.
* There is any concern by the investigator regarding the safe participation of the subject in the study or, for any other reason, the investigator considers the subject inappropriate for participation in the study.
* Patient has taken within 5 weeks of Visit 1 or anticipates a need to take oral corticosteroids during the study period except as administered per protocol.
* During Visits 2-5, there is any concern by the investigator regarding the further safe participation of the subject in the study for any reason including but not limited to history and symptoms suggestive of an impending exacerbation (e.g. a drop or downward trend in PEF from the patients personal best values) and/or noncompliance with instructions or medications.
* Patient has unresolved signs and/or symptoms of an upper respiratory tract infection or has had antibiotics administered within 4 weeks of Visit 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-01; Primary Completion 2015-09 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in VH assessed by oxygen-enhanced 1H MRI (Oe 1H MRI) after two weeks of montelukast or prednisone treatment | Baseline and after two weeks of drug treatment
Change from baseline in VH assessed by 19F-perfluoropropane MRI (19F MRI) after two weeks of montelukast or prednisone treatment | Baseline and after two weeks of drug treatment
Change from baseline in VH assessed by Lung Clearance Index (LCI) after two weeks of montelukast or prednisone treatment | Baseline and after two weeks of drug treatment
Change from baseline in VH assessed by Conducting Airway Heterogeneity (Scond) after two weeks of montelukast or prednisone treatment | Baseline and after two weeks of drug treatment
Change from baseline in VH assessed by Forced Expiratory Volume in 1 second (FEV1) after two weeks of montelukast or prednisone treatment | Baseline and after two weeks of drug treatment

SECONDARY OUTCOMES:
Comparison of VH assessed by Oe 1H MRI, 19F MRI, LCI, Scond and FEV1 at baseline | Baseline
Short-term test-retest repeatability of VH by Oe 1H MRI and 19F MRI | Visit 2 and Visit 3
Mid-term test-retest repeatability of VH by Oe 1H MRI and 19F MRI | Visit 3 and Visit 4/Visit 5

CONTACTS AND LOCATIONS:
Overall Officials: Cecil Charles, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States